CLINICAL TRIAL: NCT01636843
Title: A Randomised, Double Blind, Placebo-controlled, Multiple Dose, Phase 2b, 24 Week Trial Followed by an Open Label Extension of NNC0109-0012, an Anti-IL-20 Biologic, in Patients With Active Rheumatoid Arthritis Who Are Inadequate Responders to Methotrexate
Brief Title: A Trial of NNC0109-0012, an Anti-IL-20 Biologic, in Patients With Active Rheumatoid Arthritis Who Are Inadequate Responders to Methotrexate
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8226-3613; 2012-000610-11 (EudraCT Number); U1111-1127-9324 (Other: WHO)
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid | interventions — Fletikumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 60 mg (Experimental)
  Interventions: Drug: NNC0109-0012
- 120 mg (Experimental)
  Interventions: Drug: NNC0109-0012
- 240 mg (Experimental)
  Interventions: Drug: NNC0109-0012
- Placebo (Experimental)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0109-0012 — Administered subcutaneously (s.c., under the skin), once weekly.
  Arms: 120 mg; 240 mg; 60 mg
Drug: placebo — Administered subcutaneously (s.c., under the skin), once weekly.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe, North America and South America. The aim of this trial is to investigate the clinical efficacy of NNC0109-0012, a human monoclonal antibody, compared to placebo when administered as weekly repeat subcutaneous (under the skin) injections in to patients with active rheumatoid arthritis (RA) with inadequate responses to methotrexate (MTX) while on a stable background of MTX therapy.

ELIGIBILITY:
Inclusion Criteria: - Informed consent must be obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial - A documented diagnosis of RA at least 6 months prior to screening visit, according to the American College of Rheumatology (EULAR/ACR 2010 criteria) or by standard criteria (ACR 1987) if diagnosis was made earlier than 2010 - Active RA, characterised by: a. more than 5 tender and more than 5 swollen joints based on a 28 joint count b. C-reactive protein (CRP) above or equal to 1.0 mg/dL (10 mg/L) - Patients can be on methotrexate with or without hydroxychloroquine/chloroquine: a. Methotrexate treatment (above or equal to 15.0 mg/week) for at least 16 weeks, (above or equal to 15.0 mg/week to below or equal to 25 mg/week) for at least 8 weeks prior to screening. Patient can be on MTX as low as 10 mg/week only if due to MTX intolerance b. Hydroxychloroquine (200-400 mg/day per os, oral dosing (p.o.)) or chloroquine (250-500 mg/day p.o.) treatment for at least 8 weeks prior to screening visit Exclusion Criteria: - Patients with arthritis due to other autoimmune diseases than RA - Any active or ongoing bacterial infections within 4 weeks prior to screening visit, unless treated and resolved with appropriate therapy or any history of recurrent infections or conditions predisposing to chronic infections (e.g., bronchiectasis, chronic osteomyelitis) - History of severe, systemic viral or fungal infections within the past 6 months prior to screening visit, unless treated and/or resolved with appropriate therapy - Patients with active malignancy within the previous 5 years with the exception of adequately treated and cured basal or squamous cell carcinoma of the skin or cervical carcinoma in situ occurring more than 12 months prior to screening visit - Females of childbearing potential who are pregnant or breast feeding or intend to become pregnant - Any other disease or clinically significant abnormality in laboratory parameters which, according to the Investigator, might compromise the safety of the patient, interfere with participation in the trial or compromise the trial objective

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2012-10-30 (Actual); Primary Completion 2014-11-10 (Actual); Study Completion 2014-11-10 (Actual)

PRIMARY OUTCOMES:
ACR20 (defined as 20% improvement in American College of Rheumatology criteria measures) | At week 12 (responder or non-responder)

SECONDARY OUTCOMES:
ACR20, ACR50 and ACR70 improvement of ACR score from baseline | At weeks 12 and 24
Change in DAS28-CRP (defined as Disease Activity Score for 28 joints with C-reactive protein measure) from baseline | At weeks 12 and 24
Simplified Disease Activity Index (SDAI) remission (SDAI of 3.3 or below) | At weeks 12 and 24
European League Against Rheumatism (EULAR) criteria response | At weeks 12 and 24
Change from baseline in the overall scores of Short Form Health Survey (SF-36v2) | At weeks 12 and 24
Change from baseline in the overall scores of Health Assessment Questionnaire - Disability Index (HAQ-DI) | At weeks 12 and 24
Incidence and type of adverse events (AEs) | At weeks 12 and 24
Change from baseline in van der Heijde modified Sharp score | At weeks 12 and 24
ACR20/50/70 (20%, 50% or 70% improvement of ACR (American College of Rheumatology) score from baseline) | Week 52
Incidence and type of adverse events (AEs) | Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (114):
- United States (29):
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Placentia, California
  - Novo Nordisk Investigational Site, Upland, California
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Rock Island, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, South Bend, Indiana
  - Novo Nordisk Investigational Site, Cedar Rapids, Iowa
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Elizabethtown, Kentucky
  - Novo Nordisk Investigational Site, Lake Charles, Louisiana
  - Novo Nordisk Investigational Site, Hagerstown, Maryland
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Kalispell, Montana
  - Novo Nordisk Investigational Site, Freehold, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Lake Success, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, Orangeburg, South Carolina
  - Novo Nordisk Investigational Site, Jackson, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Mesquite, Texas
  - Novo Nordisk Investigational Site, Beckley, West Virginia
- Argentina (7):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Ciudad Autonoma Buenos Aires
  - Novo Nordisk Investigational Site, Ciudad Autonoma de Buenos Aire
  - Novo Nordisk Investigational Site, Ciudad de Buenos Aires
  - Novo Nordisk Investigational Site, Rosario
  - Novo Nordisk Investigational Site, San Juan
  - Novo Nordisk Investigational Site, San Miguel de Tucumán
- Belgium (3):
  - Novo Nordisk Investigational Site, Anderlecht
  - Novo Nordisk Investigational Site, Kortrijk
  - Novo Nordisk Investigational Site, Liège
- Brazil (9):
  - Novo Nordisk Investigational Site, Saint Oeste, Goiás
  - Novo Nordisk Investigational Site, Juiz de Fora, Minas Gerais
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Vila Clementino, São Paulo
  - Novo Nordisk Investigational Site, Cuiaba Mount
  - Novo Nordisk Investigational Site, Curitiba
  - Novo Nordisk Investigational Site, Rio de Janeiro
  - Novo Nordisk Investigational Site, São Paulo
- Czechia (5):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Hlučín
  - Novo Nordisk Investigational Site, Pardubice
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Zlín
- France (4):
  - Novo Nordisk Investigational Site, Échirolles
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Orléans
  - Novo Nordisk Investigational Site, Rennes
- Germany (7):
  - Novo Nordisk Investigational Site, Aachen
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Herne
  - Novo Nordisk Investigational Site, Koein
  - Novo Nordisk Investigational Site, Vogelsang-Gommern
- Novo Nordisk Investigational Site, Kiskunhalas, Hungary
- Italy (6):
  - Novo Nordisk Investigational Site, Arenzano
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Genova
  - Novo Nordisk Investigational Site, Iesi
  - Novo Nordisk Investigational Site, Rome
  - Novo Nordisk Investigational Site, Verona
- Mexico (10):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
  - Novo Nordisk Investigational Site, México, México, D.F.
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
  - Novo Nordisk Investigational Site, Culiacán, Sinaloa
  - Novo Nordisk Investigational Site, Chihuahua City
  - Novo Nordisk Investigational Site, Mexico City
  - Novo Nordisk Investigational Site, Monterrey N.L.
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, San Luis Potosí City
- Poland (8):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdynia
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Środa Wielkopolska
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Russia (10):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Kemerovo
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Petrozavodsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Smolensk
  - Novo Nordisk Investigational Site, Stavropol
  - Novo Nordisk Investigational Site, Yaroslavl
  - Novo Nordisk Investigational Site, Yekaterinburg
- Spain (5):
  - Novo Nordisk Investigational Site, Guadalajara
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- Ukraine (10):
  - Novo Nordisk Investigational Site, Donetsk
  - Novo Nordisk Investigational Site, Ivano-Frankivsk
  - Novo Nordisk Investigational Site, Kharkiv
  - Novo Nordisk Investigational Site, Kiev
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Luhansk
  - Novo Nordisk Investigational Site, Odesa
  - Novo Nordisk Investigational Site, Poltava
  - Novo Nordisk Investigational Site, Vinnytsia
  - Novo Nordisk Investigational Site, Zaporizhzhia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com